CLINICAL TRIAL: NCT05626738
Title: Multicenter Clinical Trial for the Evaluation of Safety and Effectiveness of Endorail in Patients With Long-lasting Colonoscopy
Brief Title: Endorail in Long Lasting Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endostart srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Endorail
Record Dates: First submitted 2022-11-08; First posted 2022-11-25 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Colonoscopy; Incomplete Colonoscopy
Keywords: Medical Device; Colonoscopy; Gastrointestinal endoscopy; Magnetic Balloon Technology; Looping; Safety; Effectiveness

STUDY DESIGN:
Intervention Model Description: Multi Centre, Post Market, Single Arm, Open-Label, Interventional Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long-lasting Colonoscopy With Endorail (Experimental): In case of long-lasting colonoscopy, Endorail is used to facilitate the completion of the procedure.
  Interventions: Device: ENDORAIL

INTERVENTIONS:
Device: ENDORAIL — In case caecal intubation time is longer than 10 minutes, the balloon catheter is inserted in the tool channel, advanced beyond the colonoscope tip and filled with Ferromagnetic Fluid. By applying the Endorail Handpiece over the patient abdomen, the balloon can be magnetically anchored. The anchored balloon guide allows to straighten the scope and the colon itself. The colonoscope can thus be easily moved back and forward along the anchored guide to facilitate colonoscope positioning and colonoscopy completion. Afterward, Endorail is removed and the straightened colonoscope can be easily pushed forward to achieve colonoscopy completion according to standard endoscopic technique.
  Other Names: Endorail Set - Endorail System

SUMMARY:
Patients with long lasting colonoscopy are characterized by higher risk of incompletion. Endorail is an accessory for colonoscopy aimed at facilitating progression of the endoscope in the large intestine. Endorail works as a magnetic anchor that is able to guide the colonoscope and to straighten colon curves and loops. The aim of this study is to test the safety and efficacy of Endorail in ensuring that incompletion rate in long-lasting colonoscopies is lower than the 10% threshold. Outpatients of either sex aged between 22-75 years undergoing elective diagnostic or surveillance colonoscopy with caecal intubation time greater than 10 minutes will take part in the study. The primary efficacy endpoint is the percentage minor or equal to 10% of incomplete long-lasting colonoscopies. The primary safety endpoints are the absence of device-related serious adverse events and the evaluation of the equality or reduction of the adverse events rates compared to diagnostic colonoscopies without Endorail.

DETAILED DESCRIPTION:
Patients with long lasting colonoscopy are characterized by higher risk of incompletion. A colonoscopy can be defined as incomplete when the endoscopist cannot reach the caecum. Caecal intubation is one of the main goals of colonoscopy and represents a diagnostic quality indicator. International guidelines recommend caecal intubation rates ≥90% for all colonoscopies in daily clinical practice. Reported incomplete colonoscopy rates range from 4% to 25%. Caecal intubation fails in 4-10% of cases in tertiary referred centres, instead in national surveys colonoscopies are incomplete in 10-25% of cases.

Endorail is a medical device intended to facilitate the positioning of a standard colonoscope. Endorail is a colonoscopy add-on device that works as a magnetic anchor able to guide the colonoscope and to straighten colon curves and loops.

Endorail is composed by the following two CE marked medical devices: Endorail Set and Endorail System. Endorail Set consists of the Endorail Balloon Guide, The Endorail Solution Syringe, The Endorail Powder and the Spike. Endorail System consists of the Endorail Handpiece and the Endorail Cart.

The aim of this study is to test the safety and efficacy of the Endorail in ensuring that incompletion rate in long-lasting colonoscopies is lower than the 10% threshold.

Outpatients of either sex aged between 22-75 years, undergoing elective colonoscopy for diagnostic or surveillance colonoscopy, who have signed a written informed consent and presenting caecal intubation time greater than 10 minutes, will take part in the study. The study plan will include a screening/baseline/treatment visit (Visit 1/Day 1), during which colonoscopy with the investigational medical device Endorail will be performed and a phone follow-up visit (Visit 2), scheduled at 7 (± 1) day after treatment with the investigational medical device Endorail.

The primary efficacy endpoint is the percentage minor or equal to 10% of incomplete long-lasting colonoscopies

The primary safety endpoints are:

* The absence of device-related serious adverse events. AND
* The evaluation of the equality or reduction of the adverse events rates compared to diagnostic colonoscopies without Endorail.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged between 22 - 75 years (inclusive);
2. Outpatients undergoing long-lasting diagnostic and surveillance colonoscopy; long-lasting colonoscopy is defined as follows: colonoscopy completion (caecal intubation) not achieved after 10 minutes from endoscope insertion through the anal canal;
3. Patients have given a written informed consent for participation in the study at the time of enrolment or before;
4. Patients able to understand the full nature and the purpose of the investigation, including possible risks and side effects, able to cooperate with the Investigator and to comply with the requirements of the entire investigation based on Investigator's judgement.

Exclusion Criteria:

1. Body mass index (BMI) > 30 kg/m2;
2. Outpatients undergoing colonoscopy for colorectal cancer screening or therapeutic indication;
3. Patients in class >2 physical status of the classification system of American Society of Anaesthesiologists;
4. Any contraindications to colonoscopy;
5. Any contraindications to sedation;
6. Known allergy or hypersensitivity to any of the elements of the Endorail Set (e.g.: iron);
7. Patients with permanently or semi-permanently implanted medical devices, (e.g. orthopedic implants, trauma fixation devices, cardiac pacemakers, implantable cardioverter defibrillator, drug pumps, neurostimulators, vascular stents, cochlear implants, aneurysm clip);
8. Presence of dense diverticulosis
9. Presence of diverticulitis
10. Presence of ferromagnetic foreign body;
11. Presence of large abdominal hernias;
12. Presence of severe thrombocytopenia;
13. Presence of severe granulocytopenia;
14. Presence of severe coagulopathy;
15. Presence of peritonitis;
16. Presence of colonic wall ischemia or necrosis or injured mucosa;
17. Presence of peritoneal carcinomatosis;
18. Boston Bowel Preparation Scale <2 in at least one of the colonic segments;
19. Presence of obstructing masses and strictures of the colon;
20. History of total or subtotal colectomy.
21. Presence of angulated and fixed colon curves;
22. Pregnant or breast-feeding women;
23. Patient unable to provide the signed informed consent, uncooperative patient or patient unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study;
24. Presence of any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromises the subject safety
25. Concomitant participation in other clinical investigations or participation in the evaluation of any investigational product/device in the 30 days before this study or previous participation in the same investigation;
26. Urgent colonoscopy.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro F Ferri, Study Director — Advice Pharma Group S.r.l.
Locations (3):
- University Hospitals, Leuven, Belgium
- Gastrozentrum, Lippe, Germany
- Humanitas, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial Initiation Date: 25 January 2023 Trial Completion Date: 25 July 2023
  Coordinating / Principal Investigator:
  * IRCCS Humanitas Research Hospital, Via Manzoni 56, I-20089 Rozzano (Milan, Italy). PI: Prof. Alessandro Repici.
  * GastroZentrum Lippe, Lange Str.55, Bad Salzuflen (Germany). PI: Prof. Helmut Neumann
  * University Hospitals Leuven. Herestraat 49, B-3000 Leuven (Belgium). PI: Prof. Raf Bisschops
Period: Overall Study
Arm/Group | Long-lasting Colonoscopy With Endorail
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients undergoing long-lasting (caecal intubation time > 10 min) diagnostic or surveillance colonoscopy
Arm/Group | Long-lasting Colonoscopy With Endorail
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 2
  Italy | 21
  Germany | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Incomplete Long-lasting Colonscopies
Description: Colonoscopy is defined completed when caecal intubation is achieved. Colonoscopy is defined long-lasting when caecal intubation time is longer than 10 minutes. The percentage of incomplete long-lasting colonscopies is calculated as the ratio, in percetange, between the number of incomplete long-lasting colonscopies and the total number of patients enrolled.
Time Frame: day 1
Measure: Number; unit: % of participants
Arm/Group | Long-lasting Colonoscopy With Endorail
Number analyzed (Participants) | 38
% of participants | 0

2. Primary Outcome: Number of Device-related Serious Adverse Events
Description: Number of the device-related serious adverse events collected at day 1 visit
Time Frame: day 1
Measure: Number; unit: Number of Device-related SAE
Arm/Group | Long-lasting Colonoscopy With Endorail
Number analyzed (Participants) | 38
Number of Device-related SAE | 0

3. Primary Outcome: Number of Device-related Serious Adverse Events
Description: Number of device-related serious adverse events collected through phone call at day 7.
Time Frame: day 7
Measure: Number; unit: Number of Device-related SAE
Arm/Group | Long-lasting Colonoscopy With Endorail
Number analyzed (Participants) | 36
Number of Device-related SAE | 0

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Long-lasting Colonoscopy With Endorail
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 2/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long-lasting Colonoscopy With Endorail (N=38)
Hypogastric pain (Gastrointestinal disorders) | 1 (1)
Hemorroidal plexus infiam-mation (Gastrointestinal disorders) | 1 (1)
Seasonal allergy (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT05626738/Prot_SAP_000.pdf